CLINICAL TRIAL: NCT01936818
Title: Study Evaluating Nasal Symptoms Induced by a Nasal Allergen Challenge (NAC) To House Dust Mite Allergen
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-100-0008
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A Multi-Center Study Evaluating the Nasal Allergic Symptomatology Induced by a Nasal Allergen Challenge (NAC) in a Dust Mite Population

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* positive ST to Dust Mite
* history of allergic rhinitis

Exclusion Criteria:

* no active infections
* no disallowed medications
* no nasal anatomical deformities or nasal surgical interventions in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects at least 18 years of age of either sex and any race
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
TNSS= total nasal symptoms score | 15 minutes

SECONDARY OUTCOMES:
Individual nasal symptoms | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ora Clinical Research Center, Andover, Massachusetts, United States